CLINICAL TRIAL: NCT07273903
Title: Subcutaneous Immunoglobulin Therapy Effectiveness Monitoring in CIDP Patients Using Smart Devices
Acronym: STEPS
Status: Not yet recruiting | Type: Observational
Sponsor: Heinrich-Heine University, Duesseldorf (Other)
Responsible Party: Principal Investigator, Dr. med. Marc Günter Pawlitzki, Study coordinator / PI, Heinrich-Heine University, Duesseldorf
Other Study IDs: STEPS_1.0
Record Dates: First submitted 2025-11-27; First posted 2025-12-10 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-11

CONDITIONS: CIDP - Chronic Inflammatory Demyelinating Polyneuropathy
Keywords: CIDP; IVIG; SCIG; wearable; steps; sleep; DHT
MeSH Terms: conditions — Polyradiculoneuropathy, Chronic Inflammatory Demyelinating

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- CIDP patients: CIDP patients (≥18 years) with typical or possible typical CIDP (2021 EAN/PNS criteria), Switched from IVIG to fSCIG within 6 months or during recruitment, Must be able to use smartwatch + smartphone, Exclude: CIDP variants, pregnancy, breastfeeding, inability to use devices

SUMMARY:
Chronic inflammatory demyelinating polyneuropathy (CIDP) is a rare autoimmune disease that affects the peripheral nerves. It causes progressive weakness and sensory loss in the arms and legs, which can severely limit daily activities. Many patients need long-term treatment with immunoglobulins, either through intravenous infusions (IVIG) or subcutaneous injections (fSCIG).

The S.T.E.P.S. study aims to explore how digital health technologies-specifically smartwatches-can help monitor the disease course and treatment effects in CIDP patients who use fSCIG at home. Current clinical tests are useful but sometimes miss small changes in strength or function. Wearables may provide a more detailed and continuous picture of patients' health between clinic visits.

Study Goals:

The main goal is to find out whether smartwatch data (such as step count and physical activity) reflect disease severity and treatment response when compared to standard clinical scores like the Inflammatory Neuropathy Cause and Treatment (INCAT) scale and the Inflammatory Rasch-built Overall Disability Scale (I-RODS).

Secondary goals include:

Assessing how smartwatch data relate to patients' quality of life and sleep patterns.

Comparing smartwatch results with other clinical scores such as muscle strength (MRC sum score) and grip strength.

Evaluating how well patients can use the smartwatch over the long term during home treatment.

An additional exploratory goal is to see whether smartwatch data can detect early signs of worsening disease before symptoms appear.

Study Design:

This is a 12-month observational study with five main clinic visits (at 0, 3, 6, 9, and 12 months). After enrolling, participants will begin or continue subcutaneous immunoglobulin therapy as decided by their treating physician. Each visit includes standard clinical assessments and questionnaires.

Participants will receive a smartwatch at the start of the study to continuously track their activity and sleep patterns. A follow-up phone call one week later will check that the device is working properly.

Duration:

Recruitment will last about 6 months, and each participant will be followed for 12 months.

Why This Matters:

By combining established clinical measures with continuous digital monitoring, the S.T.E.P.S. study may help improve understanding of disease activity and treatment response in CIDP. This could lead to more personalized therapy schedules and better long-term care for patients.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed typical or possible typical CIDP according to the 2021 EAN/PNS criteria
* Age ≥18 years
* Ability to use a smartwatch as decided by the investigator
* switched from IVIG to fSCIG within the prior 6 months or plan to switch during study recruitment phase
* on investigator-confirmed stable IVIG therapy pre-switch

Exclusion Criteria:

* Age < 18 years
* Inability to operate smartwatch or smartphone device
* current pregnancy and breastfeeding status
* CIDP variants according to the 2021 EAN/PNS criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: CIDP adult patients (≥18 years) with typical or possible typical CIDP (2021 EAN/PNS criteria), switched from IVIG to fSCIG within 6 months or during recruitment
Sampling Method: Non-Probability Sample
Enrollment: 35 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2028-01 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Change in Inflammatory Rasch-built Overall Disability Scale (I-RODS) | Baseline up to 12 months, 5 visits (months 0, 3, 6, 9, and 12)
  24-item scale, with each item representing a common, daily activity minimum value: 0 points, maximum value: 48 points, best result: 48 points
Change in Inflammatory Neuropathy Cause and Treatment (INCAT) disability score | Baseline up to 12 months, 5 visits (months 0, 3, 6, 9, and 12)
  minimum value: 0 points, maximum value: 10 points, best result: 0 points
Longitudinal development of activity parameter: step count | 365 days
Longitudinal development of activity parameter: duration of moderate activity (seconds) defined by Withings | 365 days
  Examples for moderate activity:
  Walking fast, Cleaning (vacuuming, washing windows, etc.), Playing doubles tennis or badminton, Taking a bike ride, Gardening

SECONDARY OUTCOMES:
Change in Grip strength | Baseline up to 12 months, 5 visits (months 0, 3, 6, 9, and 12)
  Measured via Vigorimeter in kPa
Change in Medical Research Council (MRC)-Sumscore | Baseline up to 12 months, 5 visits (months 0, 3, 6, 9, and 12)
  minimum value: 0 points, maximum value: 60 points, best result: 60 points
Longitudinal development of activity parameter: approximate distance traveled (meter) | 365 days
Longitudinal development of activity parameter: duration of soft activity (seconds) defined by Withings | 365 days
  Examples for soft activity:
  Sleeping, Sitting quietly, Walking slowly, Typing on a computer keyboard while seated, Watching television, Doing the dishes
Longitudinal development of activity parameter: duration of intense activity (seconds) defined by Withings | 365 days
  Examples for intense activity:
  Hiking, Running, Carrying heavy loads, Riding a bike, Playing football,baseball, or tennis (singles), Playing jump rope
Longitudinal development of activity parameter: sum of all active time (seconds) | 365 days
Wearing time of smartwatch (daily) | Baseline up to 12 months, 5 visits (months 0, 3, 6, 9, and 12)
Longitudinal development of activity parameter: approximate calories burned | Baseline up to 12 months, 5 visits (months 0, 3, 6, 9, and 12)
Change in Subjective occurrence of end-of-dose phenomena/wearing off | Baseline up to 12 months, 5 visits (months 0, 3, 6, 9, and 12)
Change in Quality of life (QoL) | Baseline up to 12 months, 5 visits (months 0, 3, 6, 9, and 12)
  The Quality of Life Questionnaire (QoL) is an instrument for measuring patients' subjective quality of life in a wide range of specific areas, WHOQOL-BREF (World Health Organization Quality of Life - abbreviated version)
Change in Pittsburgh Sleep Quality Index (PSQI) | Baseline up to 12 months, 5 visits (months 0, 3, 6, 9, and 12)
Change in Blood analysis (levels of sNfl, serum proteomics) | Baseline up to 12 months, 5 visits (months 0, 3, 6, 9, and 12)
Questionnaire about smartwatch usage | End of study visit (after 12 months, V5)
Longitudinal development of sleep parameter: time awake (seconds) | 365 days
Longitudinal development of sleep parameter: number of times user woke up | 365 days
Longitudinal development of sleep parameter: time to sleep (seconds) | 365 days
Longitudinal development of sleep parameter: total time in bed (seconds) | 365 days
Longitudinal development of sleep parameter: total time asleep (seconds) | 365 days
Longitudinal development of sleep parameter: WASO | 365 days
  Wake after sleep onset (WASO): total time asleep divided by total time in bed
Longitudinal development of sleep parameter: time spent in bed before falling asleep (seconds) | 365 days
Longitudinal development of sleep parameter: time awake after first falling asleep (seconds) | 365 days
Longitudinal development of sleep parameter: Withings Sleep score | 365 days
  Defined by Withings as follows: It measures every night's sleep and provides a score out of 100 points based on 4 key inputs:
  * Duration (total time spent sleeping)
  * Depth (part of night spent in restorative phases and deep sleep)
  * Regularity (consistency between your bed- and rise-times)
  * Interruptions (time spent awake)
Longitudinal development of cardiovascular parameter: average heartrate | 365 days
Longitudinal development of cardiovascular parameter: maximal heartrate | 365 days
Longitudinal development of cardiovascular parameter: minimum heartrate | 365
Longitudinal development of cardiovascular parameter: time in light heartrate zone (seconds) | 365 days
  Light heartrate zone is defined by Withings as follows: from 0% inclusive to 50% exclusive of maximum heart rate.
Longitudinal development of cardiovascular parameter: time in moderate heartrate zone (seconds) | 365 days
  Moderate heartrate zone is defined by Withings as follows: from 50% included to 70% excluded of maximal heart rate.
Longitudinal development of cardiovascular parameter: time in intense heartrate zone (seconds) | 365 days
  Intense heartrate zone is defined by Withings as follows: from 70% included to 90% excluded of maximal heart rate.
Longitudinal development of cardiovascular parameter: time in maximal heartrate zone (seconds) | 365 days
  Maximal heartrate zone is defined by Withings as follows: from 90% included to 100% included of maximal heart rate.
Number and time of Irregular 1-channel ECGs (according to Withings algorithm) | 365 days

CONTACTS AND LOCATIONS:
Overall Officials: Marc G Pawlitzki, PD Dr. med., Principal Investigator — Department of Neurology, Heinrich-Heine University, and University Hospital Duesseldorf, Germany
Locations (2):
- Germany (2):
  - University Hospital Düsseldorf, Düsseldorf, North Rhine-Westphalia
  - University Hospital Münster, Münster, North Rhine-Westphalia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Masanneck L, Voth J, Gmahl N, Jendretzky K, Huntemann N, Werner NM, Schmidt L, Oeztuerk M, Quint P, Schroeter CB, Hartung HP, Skripuletz T, Meyer Zu Horste G, Ruck T, Meuth SG, Pawlitzki M. Digital Activity Markers in Chronic Inflammatory Demyelinating Polyneuropathy. Ann Clin Transl Neurol. 2025 Oct;12(10):2045-2055. doi: 10.1002/acn3.70137. Epub 2025 Jul 9. PMID 40635238